CLINICAL TRIAL: NCT02400970
Title: Study About Contamination of Testicle Tissue by RT-PCR in Children With Solid Tumors
Brief Title: Contamination of Testicle Tissue by RT-PCR in Participants With Solid Tumors
Acronym: TESTIMAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0230
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Minimal Residual Disease; Fertility Preservation
Keywords: Polymerase Chain Reaction; fertility preservation
MeSH Terms: conditions — Neoplasm, Residual

INTERVENTIONS:
Other: malignant cells

SUMMARY:
For prepubertal patients, cryopreservation of testicular tissue is the only option available to preserve their fertility before cancer treatment. But testicular autograft raises the issue of the risk of reintroduction of potentially malignant cells. The aim of our study is to develop a specific and sensitive method for residual disease detection in the testicular tissue from patients treated for a solid tumor during infancy, whose fertility may have been compromised by treatments and who benefited of testicular tissue cryopreservation.

DETAILED DESCRIPTION:
Some solid tumors have high risk of metastatic localization including in testis. There is concern over the possible presence of malignant cells in testicular tissue that could cause a recurrence of the primary disease after reimplantation. Thus, the possibility of testicular tissue involvement needs to be evaluated with sensitive molecular methods.

Based on our experience in detection by RT-PCR of minimal residual disease (MRD) in neuroblastoma since 1994 [Tchirkov et al. 2003] and in testicular tissue cryopreservation since 2012, we want to develop a specific and sensitive method for residual disease detection by RT-PCR in order to evaluate the tumor contamination of testicular harvested tissue.

Study population: We chose 3 models of pediatric solid tumors with high risk of metastases and which often require sterilizing treatments (chemo and/or radiotherapy): neuroblastoma, Ewing tumor and alveolar rhabdosarcoma. We will use four tumor cells lines: IMR32 and SK-NSH for neuroblastoma; RD-ES for Ewing tumor; RH-30 for rhabdosarcoma. We plan to use 20 fragments per line.

Study duration: 12 months Study design: Testicular tissue without known malignancy but with a condition warranting a biopsy (fertility assessment) will be harvested.

The harvested testicular cortex will be treated to recover all viable sperm and then, we use remaining tissue to be contaminated with tumor cells lines. Then, detection of the specific transcript will be done by RT-PCR in fresh tissue and after freeze/thaw. Total RNA will be extracted with the TRI-reagent and qRT-PCR will be performed using the "TaqMan" technology.

Primary endpoint: to reach a sensitivity about 1/106 cells.

ELIGIBILITY:
Inclusion Criteria:

* Men in childbearing age whose fertility assessment require a testicular biopsy may be included

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients treated for a solid tumor during infancy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
malignant cells about 1/10 *6 cells. | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Justyna KANOLD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Chaput L, Greze V, Halle P, Radosevic-Robin N, Pereira B, Veronese L, Lejeune H, Durand P, Martin G, Sanfilippo S, Canis M, Kanold J, Tchirkov A, Brugnon F. Sensitive and Specific Detection of Ewing Sarcoma Minimal Residual Disease in Ovarian and Testicular Tissues in an In Vitro Model. Cancers (Basel). 2019 Nov 17;11(11):1807. doi: 10.3390/cancers11111807. PMID 31744224